CLINICAL TRIAL: NCT01635621
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Olokizumab Administered Subcutaneously to Subjects With Moderate to Severe Crohn's Disease
Brief Title: A Phase II Study to Assess the Efficacy and Safety of Olokizumab in Patients With Crohn's Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was withdrawn due to delay in timelines. There were no safety concerns regarding the study or the compound in the decision to withdraw the trial.
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CD0001; 2011-002517-11 (EudraCT Number)
Record Dates: First submitted 2012-07-03; First posted 2012-07-09 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Crohn's Disease
Keywords: Olokizumab; OKZ; CDP6038; Crohn's Disease; CDAI; IBDQ
MeSH Terms: conditions — Crohn Disease | interventions — olokizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- OKZ 120 mg (Experimental)
  Interventions: Drug: Olokizumab (OKZ)
- OKZ 240 mg (Experimental)
  Interventions: Drug: Olokizumab (OKZ)
- OKZ 120 mg with 480 mg loading dose at Week 0 (Experimental)
  Interventions: Drug: Olokizumab (OKZ)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olokizumab (OKZ) — Subjects will receive one of the following treatment regimens as subcutaneous injection solution on Weeks 0, 2, 4, 6, 8, 10, 12 and 14 of the Treatment Period:
  * OKZ 120 mg every 2 weeks
  * OKZ 240 mg every 2 weeks
  * OKZ 120 mg every 2 weeks, with a loading dose of OKZ 480 mg at Week 0
  1.6 mL of OKZ drug substance presented in a glass vial with a 1.2 mL extractable volume at a concentration of 100 mg/mL in the formulation buffer, containing 25 mM sodium citrate, 90 mM sodium chloride, 0.02 % (weight/volume) polysorbate 80, pH 6.0.
  Other Names: CDP6038
  Arms: OKZ 120 mg; OKZ 120 mg with 480 mg loading dose at Week 0; OKZ 240 mg
Drug: Placebo — Subjects will receive Placebo every 2 weeks as a subcutaneous injection solution (0.9% sodium chloride preservative-free for injection) on Weeks 0, 2, 4, 6, 8, 10, 12 and 14 of the Treatment Period.
  Arms: Placebo

SUMMARY:
The primary purpose of this multi-centre, double blind-study is to evaluate the clinical response of patients with moderate to severe Cohn's Disease (CD) following treatment with different doses and dose regimens of Olokizumab, relative to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, 18 to 65 years of age at Screening
* Diagnosis of CD (colonic localization) confirmed (at least 12 weeks prior to Screening) by either radiological or endoscopic evidence and/or histological examination
* Colonoscopy performed prior to first study medication administration (Week 0) with evidence of active CD and presence of ulceration but with no clinical suspicion of dysplasia or malignancy (colonoscopy to be performed after informed consent has been received, and all other Screening assessments have been completed)
* Moderately to severely active CD (CDAI score: 220 to 450, inclusive) at Baseline
* Female subjects must be either postmenopausal for at least 1 year, surgically incapable of childbearing, or effectively practicing an acceptable method of contraception (either oral/ parenteral /implantable hormonal contraceptives, intrauterine device or barrier and spermicide)

Exclusion Criteria:

* Subject has a diagnosis of Ulcerative Colitis or Indeterminant Colitis as determined by the investigator
* Subject has obstructive strictures with clinical evidence of partial or complete obstruction
* Subject has an active fistula (fistula secreting spontaneously or by gentle pressure)
* Subject has a history of diverticulitis or symptomatic diverticulosis
* Subject has any prior exposure to anti-IL-6 agents (eg, Tocilizumab)
* Female subjects who are breastfeeding, pregnant, or plan to become pregnant during the study or within 24 weeks following the last dose of the study drug
* Subject has a high risk of infection (eg, subjects with leg ulcers, indwelling urinary catheter, persistent or recurrent chest infections, and subjects who are permanently bedridden or wheelchair bound)
* Subject has a concurrent malignancy or a history of malignancy. Subjects who have been successfully treated and who have remained malignancy-free for at least 5 years prior to Screening may be included

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with clinical response or remission as measured by the Crohn's Disease Activity Index (CDAI) at Week 8 | Week 8

SECONDARY OUTCOMES:
Percentage of subjects with clinical response as measured by the Crohn's Disease Activity Index (CDAI) at Week 16 | Week 16
Percentage of subjects with clinical remission as measured by the Crohn's Disease Activity Index (CDAI) at Week 16 | Week 16
Change from Baseline in the Crohn's Disease Activity Index (CDAI) to Week 16 | From Baseline to Week 16
Change from Baseline in the Inflammatory Bowel Disease Questionnaire (IBDQ) total score at Week 16 | From Baseline to Week 16
Percentage of subjects with Inflammatory Bowel Disease Questionnaire (IBDQ) response at Week 16 | Week 16
Percentage of subjects in Inflammatory Bowel Disease Questionnaire (IBDQ) remission at Week 16 | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)